CLINICAL TRIAL: NCT03542201
Title: Comparison of Blogshot Formats With Standard Cochrane Plain Language Formats: Randomized Controlled Trial
Brief Title: Comparison of Blogshot Formats With Standard Cochrane Plain Language Formats
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IP-2014-09-7672
Record Dates: First submitted 2018-05-17; First posted 2018-05-31 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-05

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLS (Experimental): Plain abstract about the Cochrane systematic review.
  Interventions: Other: PLS
- Blogshot (Experimental): Blogshot presentation of the results of Cochrane systematic review.
  Interventions: Other: Blogshot

INTERVENTIONS:
Other: PLS — Participants will have to read standard textual information about the conducted systematic review (approximately 500 words)
  Arms: PLS
Other: Blogshot — Participants will have to read the blogshot information about the results of the Cochrane systematic review (approximately 100 words)
  Arms: Blogshot

SUMMARY:
Participants will receive in random order on format of brief description of systematic review summary on health intervention. One group will receive standard plain language summary, while another will receive Cochrane blog shot, containing only few information about the efficacy of the intervention. After reading, their task will be to answer several questions about the material they have read.

ELIGIBILITY:
Inclusion Criteria:

* Patients visiting their family doctor, students of biomedical studies.

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Understanding | 3 months
  Number of the correct answers about the content of the summary, which will consist of four multiple choice questions (with four possible answers where only one is correct, for each question) about the text the participants are reading. Questions will be developed by research team and revised by expert in health communication. The scale ranges from 0-4, where greater score indicates better understanding of the material.

SECONDARY OUTCOMES:
Reading experience | 3 months
  Likert type scale 1-10 (1 indicating low preference for current presentation type, 10 indicating absolute preference for the current presentation type.
Health numeracy | 3 months
  5 questions about the numerical tasks placed in medical content, total score is number of correct answers on those questions. The five questions are part of Numeracy Understanding in Medicine Instrument (Schapira et al, 2012), and we will translate only the questions focusing on Probability section. Cronbach's alpha in previous research was 0.86 (Schapira et al, 2012). The questions will be revised by independent translator and back translated to English.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Buljan, MPsy, Principal Investigator — PhD student
Locations (1):
- University of Split School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schapira MM, Walker CM, Cappaert KJ, Ganschow PS, Fletcher KE, McGinley EL, Del Pozo S, Schauer C, Tarima S, Jacobs EA. The numeracy understanding in medicine instrument: a measure of health numeracy developed using item response theory. Med Decis Making. 2012 Nov-Dec;32(6):851-65. doi: 10.1177/0272989X12447239. Epub 2012 May 25. PMID 22635285
- [Derived] Buljan I, Tokalic R, Roguljic M, Zakarija-Grkovic I, Vrdoljak D, Milic P, Puljak L, Marusic A. Comparison of blogshots with plain language summaries of Cochrane systematic reviews: a qualitative study and randomized trial. Trials. 2020 May 25;21(1):426. doi: 10.1186/s13063-020-04360-9. PMID 32450904